CLINICAL TRIAL: NCT02397239
Title: Comparison of Cost-effectiveness of Continuation Maintenance Therapy With Six Cycles of Pemetrexed Versus Pemetrexed Until Disease Progression for Metastatic Non-squamous Non-small-cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-BR-103-062; MOHW103-TD-B-111-06 (Other Grant/Funding Number: The Ministry of Health and Welfare, Taiwan); MOHW103-TDU-B-211-113002 (Other Grant/Funding Number: The Ministry of Health and Welfare, Taiwan)
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood hemoglobin, white blood cell, absolute neutrophil count, platelet count, total bilirubin, aspartate aminotransferase, alanine aminotransferase, creatinine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Six cycles: Maintenance pemetrexed 500 mg/m2 every 3 weeks for six cycles
- Until disease progression: Maintenance pemetrexed 500 mg/m2 every 3 weeks until disease progression

SUMMARY:
Protocol title:

Comparison of cost-effectiveness of continuation maintenance therapy with six cycles of pemetrexed versus pemetrexed until disease progression for metastatic non-squamous non-small-cell lung cancer (NSCLC)

Study design:

An open-labelled, randomized, phase 2 trial

Indication:

Patients with stage IV non-squamous NSCLC, an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, and have received first-line or second-line chemotherapy with pemetrexed plus platinum for 4 cycles

Treatment:

Maintenance pemetrexed 500 mg/m2 every 3 weeks for six cycles versus until disease progression

Objectives:

Primary endpoint:

1. Progression-free survival in the intention-to-treat population

Secondary endpoints:

1. Cost-effectiveness
2. Overall survival
3. Quality-of-life (QoL)
4. Quality-adjusted progression-free survival (QA-PFS)
5. Quality-adjusted life expectancy (QALE)
6. Tumor response rate
7. Adverse events

Planned sample size:

36 patients in each arm; total 72 patients

Total number of sites:

1 site

Duration of patient enrollment:

3 years

DETAILED DESCRIPTION:
Inclusion criteria:

1. Males and females ≥ 20 years of age
2. ECOG performance status of 0-1
3. Histologically or cytologically verified non-squamous NSCLC
4. Stage IV disease, as defined by American Joint Committee on Cancer 7th edition staging, prior to first-line or second-line chemotherapy with pemetrexed plus platinum
5. At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
6. Completion of 4 cycles of first-line or second-line chemotherapy with pemetrexed plus platinum and documented radiographic evidence of a complete or partial tumor response or stable disease by RECIST 1.1
7. Adequate organ function, including followings:

   Bone marrow:

   Absolute neutrophil count ≥ 1.5 x 103 /μL White blood cell ≥ 3.0 x 103 /μL Platelet count ≥ 75 x 103 /μL Hemoglobin ≥ 8.0 g/dL

   Hepatic:

   Total bilirubin ≤ 1.5 x upper normal limit (UNL) Aspartate aminotransferase (AST) ≤ 3.0 x UNL (≤ 5.0 x UNL if liver metastasis) Alanine aminotransferase (ALT) ≤ 3.0 x UNL (≤ 5.0 x UNL if liver metastasis)

   Renal:

   Estimated glomerular filtration rate ≥ 30 mL/min
8. Estimated life expectancy of at least 6 months
9. Ability to comply with study and follow-up procedures
10. Signed informed consent document

Exclusion criteria:

1. Squamous cell and/or mixed small-cell, non-small-cell histology
2. Prior participation in any investigational drug study within 4 weeks
3. Prior malignancy other than NSCLC, except those remain disease-free for ≥ 3 years after curative treatment, non-melanoma skin cancer or in situ cervical cancer
4. Serious concomitant systemic disorders, such as acute or recent myocardial infarction (< 6 months before enrollment), congestive heart failure with New York Heart Association functional class II~IV, frequent exacerbations of chronic obstructive pulmonary disease (≥ 2 hospitalizations per year), or recent cerebrovascular disease (< 6 months before enrollment)
5. Active uncontrolled infections or HIV infection
6. Current or planned pregnancy, or breast feeding in women
7. Symptomatic central nervous system metastasis unless the patient has completed successful local therapy and has been off corticosteroids for ≥ 4 weeks
8. Concurrent administration of any other antitumor therapy including chemotherapy, target therapy, immunotherapy, and hormone therapy
9. Psychiatric disorders that would compromise the patient's compliance or decision

Criteria for evaluation:

QoL:

QoL will be measured using the EuroQol 5-dimensional questionnaire (EQ-5D), World Health Organization Quality-of-Life, brief version (WHOQOL-BREF), European Organization for Research and Treatment of Cancer (EORTC) questionnaires.

Efficacy:

Tumor response rate will be determined by RECIST 1.1. Data of progression-free survival and overall survival will be collected for all subjects.

QA-PFS and QALE:

Investigators will adjust the progression-free survival by the utility values of QoL measured from the EQ-5D to obtain the QA-PFS. In addition, investigators will extrapolate the survival function to lifetime based on the survival ratios between patients and age- and sex-matched referents simulated from the life tables of Taiwan. After adjusting the lifetime survival by the utility values of QoL, the QALE will also be estimated using quality-adjusted life-year (QALY) as the unit.

Cost-effectiveness:

The monthly healthcare expenditures, which included National Health Insurance-reimbursed and out-of-pocket direct medical costs, will be obtained from the reimbursement database of National Cheng Kung University Hospital. These values were multiplied by the corresponding survival probabilities to calculate the lifetime costs or costs during the progression-free period. Hence, costs/life-year or costs/QALY can be obtained for comparison of cost-effectiveness.

Adverse events:

Safety parameters include laboratory adverse events (e.g., anemia, leukopenia, neutropenia, thrombocytopenia, creatinine, AST, ALT) and non-laboratory adverse events (e.g., fatigue, nausea, vomiting, mucositis/stomatitis, anorexia, diarrhea, constipation, infection, febrile neutropenia, pain, sensory neuropathy, rash, edema, watery eye). Common Terminology Criteria for Adverse Events (CTCAE) v4.0 will be used to grade toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 20 years of age
2. ECOG performance status of 0-1
3. Histologically or cytologically verified non-squamous NSCLC
4. Stage IV disease, as defined by American Joint Committee on Cancer 7th edition staging, prior to first-line or second-line chemotherapy with pemetrexed plus platinum
5. At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
6. Completion of 4 cycles of first-line or second-line chemotherapy with pemetrexed plus platinum and documented radiographic evidence of a complete or partial tumor response or stable disease by RECIST 1.1
7. Adequate organ function, including followings:

   Bone marrow:

   Absolute neutrophil count ≥ 1.5 x 103 /μL White blood cell ≥ 3.0 x 103 /μL Platelet count ≥ 75 x 103 /μL Hemoglobin ≥ 8.0 g/dL

   Hepatic:

   Total bilirubin ≤ 1.5 x upper normal limit (UNL) Aspartate aminotransferase (AST) ≤ 3.0 x UNL (≤ 5.0 x UNL if liver metastasis) Alanine aminotransferase (ALT) ≤ 3.0 x UNL (≤ 5.0 x UNL if liver metastasis)

   Renal:

   Estimated glomerular filtration rate ≥ 30 mL/min
8. Estimated life expectancy of at least 6 months
9. Ability to comply with study and follow-up procedures
10. Signed informed consent document

Exclusion Criteria:

1. Squamous cell and/or mixed small-cell, non-small-cell histology
2. Prior participation in any investigational drug study within 4 weeks
3. Prior malignancy other than NSCLC, except those remain disease-free for ≥ 3 years after curative treatment, non-melanoma skin cancer or in situ cervical cancer
4. Serious concomitant systemic disorders, such as acute or recent myocardial infarction (< 6 months before enrollment), congestive heart failure with New York Heart Association functional class II~IV, frequent exacerbations of chronic obstructive pulmonary disease (≥ 2 hospitalizations per year), or recent cerebrovascular disease (< 6 months before enrollment)
5. Active uncontrolled infections or HIV infection
6. Current or planned pregnancy, or breast feeding in women
7. Symptomatic central nervous system metastasis unless the patient has completed successful local therapy and has been off corticosteroids for ≥ 4 weeks
8. Concurrent administration of any other antitumor therapy including chemotherapy, target therapy, immunotherapy, and hormone therapy
9. Psychiatric disorders that would compromise the patient's compliance or decision

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic non-squamous mon-small-cell lung cancer
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year

SECONDARY OUTCOMES:
Cost-effectiveness: Cost/QA-PFS | 2 years
  Quality-adjusted progression-free survival (QA-PFS)
Overall survival | 1 year
Quality-of-life (QoL) Questionnaire | 1 year
Quality-adjusted progression-free survival (QA-PFS) | 1 year
Quality-adjusted life expectancy (QALE) | 1 year
Tumor response rate | 1 year
Number of Adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan